CLINICAL TRIAL: NCT00940368
Title: A Study to Evaluate the Anti-Emetic Effect of Ginger Powder Vs Placebo as an Add-on Therapy in Children and Adolescents Receiving Chemotherapy : A Randomized Controlled Trial
Brief Title: A Study to Assess the Anti-Emetic Efficacy of Ginger in Children and Adolescents Receiving Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Anu K, AIIMS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: T-10/27.02.2009
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Nausea; Vomiting
Keywords: Nausea; Vomiting; Chemotherapy
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginger arm (Experimental): The patients in this arm will be randomly selected in each cycle of chemotherapy. The unit of randomization is the cycle of chemotherapy. In each cycle of chemotherapy of all patients recruited in the study will be categorized using the computer generated random numbers. The patients in the ginger arm; Group A will be getting ginger powder capsules according to their body weight;ie;there are two weight categories within Group A:
  Category 1- 20kg-40kg Category 2- 40kg-60kg Category 1 will receive 2 capsules 3 times a day,ie; 1gram ginger powder per day Category 2 will receive 5 capsule divided in 3 doses per day,ie; 2gram ginger powder per day
  Interventions: Dietary Supplement: Provision of capsules containing ginger powder or placebo
- Placebo arm (Placebo Comparator): Patients (children and adolescents) will be included in this arm after randomization of the cycle of chemotherapy of the patient. Starch powder/Glucose powder is used as placebo.The patients in the placebo arm; Group B will be getting ginger powder capsules according to their body weight;ie;there are two weight categories within Group B:
  Category 1- 20kg-40kg Category 2- 40kg-60kg Category 1 will receive 2 capsules 3 times a day,ie; 1gram placebo powder per day Category 2 will receive 5 capsule divided in 3 doses per day,ie; 2gram placebo powder per day
  Interventions: Dietary Supplement: Provision of capsules containing ginger powder or placebo

INTERVENTIONS:
Dietary Supplement: Provision of capsules containing ginger powder or placebo — The patients(children and adolescents) will be provided with Capsules containing either ginger powder or placebo on the three days when they receive chemotherapy.
  For weight category 1(20-40kg),6 capsules are given in three divided doses and the amount of ginger powder administered per day is 1 gram.
  For weight category 2(40-60kg), 5 capsules are given in three divided doses and the amount of ginger powder administered per day is 2 gram.
  Other Names: Tulsi Ayurvedic Products & Research(P)LTd,U.P.,India

SUMMARY:
Ginger root powder is found to be significantly effective,when given as an add-on therapy in reducing chemotherapy induced nausea and vomiting in children and adolescents receiving chemotherapy.

It is very cost effective and as compared to the other add-on therapy drug like aprepitant.

DETAILED DESCRIPTION:
Cisplatin is a chemotherapeutic agent with high emetogenic potential. High doses of Cisplatin (120 mg/m2) induces nausea and vomiting in 90 % of patients. More than 60% of patients experience nausea and vomiting even if they are getting the conventional anti emetic medications.

Children and adolescents with cancer are using complementary and alternative medicine (CAM) to relieve symptoms, reduce side effects of treatment, and cope with the emotional aspects of having a life-threatening illness. Parental decisions about using CAM should be based on studies of efficacy and safety .

Ginger is already used in traditional folk medicine to treat nausea and vomiting.Additionally, ginger's ability to block 5-HT3 receptors and its free-radical scavenging action in the gut suggests that it may be beneficial for reducing both the prevalence and severity of chemotherapy induced nausea and vomiting.

Ginger is an easily available and cost effective substance in Indian scenario; (1gm costs less than one rupees). A dose of 1-2 gm of ginger is found to have favourable effects in reducing the incidence of nausea and vomiting. There are not much side-effects of ginger have been established so far, except mild stomach upset, increased burping and nausea seen in very few patients after the ingestion of ginger. Ginger is a widely available,affordable and acceptable natural substance which is to be included as an additional treatment option for chemotherapy induced nausea and vomiting which will significantly improve the health, compliance with treatment and quality of life of patients receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a histologically confirmed diagnosis of Osteosarcoma/ Malignant Fibrohistiocytoma of bone that is currently being treated with chemotherapy with high emetogenic potential chemotherapeutic agent(Cisplatin at a dose 120mg/m2 ; Adriamycin 75 mg/m2)
* Age group : 8-21 yrs.
* Weight : greater than or equal to 20 kg and less than 40 kg in Category 1
* Weight : greater than or equal to 40 kg and less than 60 kg in Category 2
* Patients who are willing to participate in study.
* Patients or their parents who can understand Hindi or English.

Exclusion Criteria:

* Patients of age <8 yrs or age >21 yrs.
* Weight < 20 kg and greater than or equal to 40 kg in Category 1
* Weight < 40 kg and greater than or equal to 60 kg in Category 2
* Patients receiving chemotherapy with drugs other than Cisplatin.
* Patients receiving a dosage of chemotherapy with Cisplatin<120 mg/m2.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-12 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in the Incidence and Severity of Chemotherapy Induced Nausea and Vomiting | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anu K, BSc.Nursing, Principal Investigator — All India Institute of Medical Sciences; Kamlesh K Sharma, MSc.Nursing, Study Director — All India Institute of Medical Sciences; Sameer Bakhshi, MD, Study Chair — All India Institute of Medical Sciences; Y K Gupta, MD,FAMS,FIPS, Study Chair — All India Institute of Medical Sciences
Locations (1):
- Dr. B.R. Ambedkar Institute Rotary Cancer Hospital, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Pillai AK, Sharma KK, Gupta YK, Bakhshi S. Anti-emetic effect of ginger powder versus placebo as an add-on therapy in children and young adults receiving high emetogenic chemotherapy. Pediatr Blood Cancer. 2011 Feb;56(2):234-8. doi: 10.1002/pbc.22778. Epub 2010 Sep 14. PMID 20842754